CLINICAL TRIAL: NCT06293768
Title: The Technological Challenge of Continuous Wireless Monitoring for the Management of Complex Patients in the Internal Medicine Departments: the "Green Line" From the Hospital to the Territory. Randomized Controlled Trial GreenLine H-T."
Brief Title: Continuous Wireless Monitoring for Patients in the Internal Medicine UOC. Randomized Controlled Trial (GreenLineH-T)
Acronym: GreenLineH-T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fadoi Foundation, Italy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: FADOI.05.2018
Record Dates: First submitted 2022-02-10; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Hospitalization
Keywords: Telemonitoring; Internal Medicine

STUDY DESIGN:
Intervention Model Description: The study involves the enrollment of 300 patients (150 patients undergoing continuous monitoring and 150 as a control). 50 of the patients undergoing continuous monitoring come from the group A and 100 from group B, same ratio in the control group.
  Group A includes patients admitted to the acute ward who are considered transferable to the ward for subacute by the seventh day of hospitalization. Group B includes patients admitted to the acute ward who are considered dismissible by the seventh day of hospitalization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A continuous monitoring (Experimental): Group A includes patients admitted to the acute ward who are considered transferable to the ward for subacute by the seventh day of hospitalization. These patients receive continuous telemonitoring of the patient's clinical condition for 5 days after transfer to the subacute ward
  Interventions: Device: continuous wireless monitoring system of Vital Signs (Win@Hospital) + continuous system for continuous monitoring of blood sugar (Dexcom G6)(only for diabetic patients)
- Group A standard monitoring (No Intervention): Group A includes patients admitted to the acute ward who are considered transferable to the ward for subacute by the seventh day of hospitalization. These patients receive standard telemonitoring of the patient's clinical condition for 5 days after transfer to the subacute ward
- Group B continuous monitoring (Experimental): Group B includes patients admitted to the acute ward who are considered dismissible by the seventh day of hospitalization. These patients receive continuous telemonitoring of the patient's clinical condition for 5 days after discharge to the home
  Interventions: Device: continuous wireless monitoring system of Vital Signs (Win@Hospital) + continuous system for continuous monitoring of blood sugar (Dexcom G6)(only for diabetic patients)
- Group B standard monitoring (No Intervention): Group B includes patients admitted to the acute ward who are considered dismissible by the seventh day of hospitalization. These patients receive standard telemonitoring of the patient's clinical condition for 5 days after discharge to the home

INTERVENTIONS:
Device: continuous wireless monitoring system of Vital Signs (Win@Hospital) + continuous system for continuous monitoring of blood sugar (Dexcom G6)(only for diabetic patients) — Patients randomized to the experimental group on discharge or with transfer to the subacute ward will be connected to the system continuous monitoring of Vital Signs(Win@Hospital) continuous system for the continuous monitoring of blood sugar(Dexcom G6)(only for diabetic patients). The system, once applied, does not require the presence of a dedicated person and continuous monitoring in real time. It is set with alerts that are triggered both when the parameters they leave the normal ranges both if the data is not recorded due to technical problems. the data is transmitted in real time on mobile devices in the possession of a doctor and a nurse available 24 hours a day who guarantee the remote control system. Devices. Mobiles also contain the clinical information of each patient.
  Arms: Group A continuous monitoring; Group B continuous monitoring

SUMMARY:
Monocentric prospective controlled randomized in open-label study. The study involves the enrollment of 300 patients (150 patients undergoing continuous monitoring and 150 as a control), aim of the study is to evaluate in these patients the efficacy of a continuous telemonitoring of the patient's clinical condition for 5 days compared to a traditional clinical monitoring.

DETAILED DESCRIPTION:
FADOI Foundation (Italian Scientific Society of Internal Medicine) has promoted a study in collaboration with the ASL Roma 6, monocentric prospective controlled randomized in open-label in patients admitted to an Internal Medicine Unit and subsequently sent to the subacute or discharged care unit. Specifically, the recruitment will take place in the Internal Medicine of the Albano Hospital - Polo H2 of the ASL Roma 6. The aim of the study is to evaluate in these patients the efficacy of a continuous telemonitoring of the patient's clinical condition for 5 days compared to a traditional clinical monitoring. 50 of the patients undergoing continuous monitoring come from the A group and 100 from group B, same ratio in the control patient group. In fact, the study consists of two patient settings, Group A and Group B. Group A includes patients admitted to the acute ward who are considered transferable to the ward for subacute by the seventh day of hospitalization. Group B includes patients admitted to the acute ward who are considered dismissible by the seventh day of hospitalization

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients discharged consecutively from the Internal Medicine Unit or transferred to the subacute ward within 7 days of hospitalization, with Blaylock Risk Assessment Screening (BRASS) ≥ 11 and at least two active pathologies
* Patients discharged consecutively from the UOC Internal Medicine or transferred to the ward of subacute within 7 days of hospitalization, with at least two active pathologies
* Signature of informed consent

Exclusion Criteria:

* Patients from RSA and Long-term care
* Terminal cancer patient
* Patients with severe cognitive disability or otherwise unable to tolerate the device
* Patients unable to express valid consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
difference in the incidence of major complications at 30 days | 30 days
  difference in the number of major complications at 30 days after transfer from the UOC for acute to that for subacute and from the hospital to the home among patients undergoing continuous remote monitoring and those subject to standard monitoring.

SECONDARY OUTCOMES:
number of acute patients who in seven days reach the criteria to be discharged or ransferred to the subacute ward | 7 days
  Percentage of patients admitted to Acute Internal Medicine who reach the criteria of transfer to the ward for subacute at 7 days and percentage of patients admitted to Internal Medicine for acute patients who reach the criteria for discharge at home at 7 days
Difference in the incidence of major complications at the end of the telemonitoring phase | 7 days
  Difference in the number of major complications at the end of the telemonitoring phase
  / standard clinical monitoring after transfer from acute to subacute UOC and from the hospital to the home between patients undergoing continuous telemonitoring and those undergoing standard monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Fontanella, MD, Study Director — FADOI FOUNDATION
Locations (1):
- Ospedale di Albano - Polo H2, Roma, Italy

IPD SHARING:
Plan to Share IPD: No